CLINICAL TRIAL: NCT01558167
Title: A phaseI/II Safety and Efficacy Trial of a Combination of Bendamustine, Rituximab and Lenalidomide (BRL) in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: A Safety and Efficacy Trial of a Combination of Bendamustine, Rituximab and Lenalidomide in Patients With Chronic Lymphocytic Leukemia
Acronym: CLL2P
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Mundipharma Research GmbH & Co KG (Industry); Roche Pharma AG (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2P; 2009-012957-39 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2012-03-20 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Dose limiting toxicity of Lenalidomide; Chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine, Rituximab,Lenalidomide (Experimental): Dose modification treatment plan of lenalidomide
  Interventions: Drug: Bendamustine, Rituximab, Lenalidomide

INTERVENTIONS:
Drug: Bendamustine, Rituximab, Lenalidomide — Bendamustine: 50 mg/m2, i.v., day 1+2
  Rituximab: Cycle 1: 375 mg/m2, i.v. day 0; Cycle 2-6: 500mg/m2, i.v., day 1
  Lenalidomide:
  * Dose level 1: Cycle 1-6: 2,5mg p.o., d1-28
  * Dose level 2: Cycle 1: 2,5mg p.o., d1-28; Cycle 2-6: 5mg p.o., d1-28
  * Dose level 3: Cycle 1: 2,5mg p.o., d1-28; Cycle 2:5mg p.o., d1-28; Cycle 3-6: 10 mg p.o., d1-28
  * Dose level 4: Cycle 1: 2,5mg p.o., d1-28; Cycle 2:5mg p.o., d1-28; Cycle 3: 10 mg p.o.,d1-28, Cycle 4-6: 15 mg p.o.,d1-28
  * Dose level 5: maximal tolerated dose
  Other Names: Ribomustine; MabThera; Revlimid

SUMMARY:
This is a prospective, multicenter, open label, non-randomized, phase I/II-study to define safety and efficacy of BRL combination in relapsed/refractory patients and to recommend a safe and efficacious dose for future phase II/III study.

Hypothesis: The simultaneous administration of BRL in relapsed CLL is feasible, safe and efficient.

DETAILED DESCRIPTION:
As too its mechanism of action lenalidomide seems to work rather by immunomodulation than by a direct anti-proliferative activity against CLL cells. Lenalidomide stimulates T- and NK-cells, modulates the tumour microenvironment in CLL and inhibits bone marrow angiogenesis. There is a rationale to combine lenalidomide with the alpha-CD20 mAb rituximab because lenalidomide enhances NK cell mediated antibody dependent cytotoxicity of rituximab treated NHL cells. On the other hand, there is increasing evidence that the combination of chemotherapy (FC) and rituximab results in highest response rates and longest progression-free survival in treatment naive and relapsed CLL. Besides FCR the combination of bendamustine, a hybrid alkylating agent with properties of a purine-analogue, with rituximab (BR) seems to be very active in relapsed and treatment-naive CLL based on results of a phase II trial of the GCLLSG. Preliminary results with lenalidomide showed a promising response rate of 32% including high risk patients. Thus, the combination of BRL could improve the therapeutic activity in high risk CLL by combining two immunomodulatory with a classic cytotoxic principle.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. 18 years of age or older.
3. Medically fit patients without relevant comorbidity, defined as total CIRS score ≤ 6.
4. WHO performance status of 0-2.
5. Confirmed diagnosis of CLL in need of treatment (Binet C or A/B with active disease) according to the updated IWCLL guidelines (Hallek et al. 2008).
6. Life expectancy > 12 weeks.
7. Relapsed or refractory disease after at least one, but no more than 3 prior regimens. Patients who previously received bendamustine (with or without rituximab) must have had at least a partial response with duration of response of at least six months.
8. CLL therapy, major surgery, or irradiation for CLL was completed > 4 weeks before registration in this study. Patients must have recovered from the acute side effects incurred as a result of previous therapy.
9. Patient is able and willing to receive adequate anticoagulation as specified in this protocol.
10. Adequate liver function as indicated by a total bilirubin, AST, and ALT ≤2 the institutional ULN value, unless directly attributable to the patient's tumor.
11. Creatinine clearance >60ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured after 24h-urine collection.
12. ANC > 1500/µl and platelet count > 75.000/μl, unless decrease is due to bone marrow involvement of CLL
13. Negative serological hepatitis B test, negative testing of hepatitis C RNA, negative HIV test within 6 weeks prior to registration.
14. Females of childbearing potential (FOCP) must understand that the study medication has a teratogenic risk and must agree to use, and be able to comply with effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 6 months after the end of study drug therapy, even if she has amenorrhea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis.

Exclusion Criteria:

1. Previously treated with > 3 prior regimens for CLL.
2. Known central nervous system (CNS) involvement of CLL.
3. Patients who have progressed with more aggressive B-cell cancers such as Richter's syndrome or are diagnosed with B-PLL.
4. History of anaphylaxis following exposure to any of the used study-drugs and/or thalidomide.
5. Evidence of TLS per the Cairo-Bishop definition of laboratory TLS (subjects may be enrolled upon correction of electrolyte abnormalities).
6. Participation in another clinical trial and/or use of investigational agents or concurrent anti cancer treatment within the last 4 weeks of registration.
7. Other severe, concurrent diseases, including tuberculosis, mental disorders, serious cardiac functional capacity (class III or IV as defined by the New York Heart Association Classification), severe diabetes, severe hypertension, pulmonary disease (COPD with hypoxemia), or major organ malfunction that could interfere with the patient's ability to participate in the study.
8. Pregnant or lactating women.
9. Any circumstance at the time of study entry that would preclude completion of the study or the required follow-up.
10. Active secondary malignancy requiring treatment (except basal cell carcinoma or malignant tumor curatively treated by surgery) within the last 5 years before registration.
11. Active bacterial, viral or fungal infection.
12. Medical condition requiring prolonged use of oral corticosteroids (> 1 month).
13. Cerebral dysfunction, legal incapacity.
14. Patients with contraindications according to Summary of Product Characteristics or Investigator's Brochure.
15. Patients who are employees of the Sponsor (University of Cologne) or the study sites.
16. Persons placed in an institution by legal or official order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
dose limiting toxicity | After 28 days of dosing at the respective target dose level of lenalidomide
  DLT defined as
  * absolute neutrophil count < 500/µl for 7 consecutive days or more
  * febrile neutropenia
  * platelet count < 20.000/µl
  * grade 4 tumour flare
  * grade 4 non-hematologic toxicity

SECONDARY OUTCOMES:
Response rate | up to 4 years
  response will be evaluated according to criteria of the CLL-Guidelines on CLL of the IWCLL-working Group.
progression free survival | up to 4 years
  Progression-free survival based on investigator's assessment:
  PFS is defined as the time from registration to the first occurrence of progression, relapse or death from any cause. Disease progression will be assessed by the investigators using the IWCLL criteria.
Overall Survival | up to 4 years
  Overall survival is defined as the time from registration to death.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, Prof.Dr., Study Chair — German CLL Study Group; Clemens Wendtner, Prof.Dr., Study Director — German CLL Study Group
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maurer C, Pflug N, Bahlo J, Kluth S, Rhein C, Cramer P, Gross-Ophoff C, Langerbeins P, Fink AM, Eichhorst B, Kreuzer KA, Fischer N, Tausch E, Stilgenbauer S, Bottcher S, Dohner H, Kneba M, Dreyling M, Binder M, Hallek M, Wendtner CM, Bergmann M, Fischer K; German CLL Study Group. Bendamustine and rituximab in combination with lenalidomide in patients with chronic lymphocytic leukemia. Eur J Haematol. 2016 Sep;97(3):253-60. doi: 10.1111/ejh.12714. Epub 2016 Feb 9. PMID 26643449